CLINICAL TRIAL: NCT06865378
Title: The Correlation Between Intraoperative End Tidal Carbon Dioxide, Perfusion Index and Pulse Variability Index on Postoperative Nausea Vomiting and Pain; Prospective Study
Brief Title: The Correlation Between Intraoperative End Tidal Carbon Dioxide, Perfusion Index and Pulse Variability Index on Postoperative Nausea Vomiting and Pain
Status: Enrolling by invitation | Type: Observational
Sponsor: Naime Yalçın (Other)
Responsible Party: Sponsor-Investigator, Naime Yalçın, Specialist Anesthesiology and Reanimation, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Other Study IDs: KAEK/2021.02.62
Record Dates: First submitted 2025-02-20; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Nausea and Vomiting; Postoperative Pain, Acute; End Tidal Carbon Dioxide; Perfusion Index and Pleth Variability Index
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Carbon Dioxide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Arm Hypocarbia
  Interventions: Procedure: Carbon dioxide (CO2) gas insufflation
- Arm normocarbia
  Interventions: Procedure: Carbon dioxide (CO2) gas insufflation
- Arm hypercarbia
  Interventions: Procedure: Carbon dioxide (CO2) gas insufflation

INTERVENTIONS:
Procedure: Carbon dioxide (CO2) gas insufflation — Artificial pneumoperitoneum created by the Trendelenburg position and carbon dioxide (CO2) insufflation, which is widely used in laparoscopic procedures, frequently leads to physiological changes such as postoperative nausea and vomiting (PONV) and pain. Therefore, the currently limited usable parameters PI and PVI will be evaluated in correlation with end tidal CO2 in continuous monitoring.

SUMMARY:
Postoperative pain, which is frequently encountered in laparoscopic operations, has been examined in different studies with end tidal CO2 (end tidal carbon dioxide), total insufflated gas amount and PI (Perfusion index) parameters. PONV (postoperative nausea and vomiting), which is encountered more frequently than pain in the postoperative period, has been examined in relation to end tidal CO2. In this study, it was aimed to evaluate the development of postoperative pain and PONV, which affect recovery and patient comfort, by comparing the relationship between end tidal CO2, PI and PVI (Pulse variability index).

DETAILED DESCRIPTION:
In recent years, laparoscopic gynecologic surgery has become a preferred technique over traditional open surgery due to its benefits such as better cosmetic results, lower risk of bleeding, minimally invasive surgery, lower postoperative pain and incidence of wound infection, and as a result, earlier discharge.

PI (Perfusion index), the ratio of alternating current component to direct current component, is a representation of the photoplethysmography waveform that quantitatively reflects real-time changes in peripheral blood flow in the monitored region. PVI (Pulse variability index) is another dynamic index and many studies have concluded that it is useful in assessing fluid responsiveness in patients. However, there are still uncertainties in the study regarding the effect of pneumoperitoneum on PVI. PVI, calculated from respiratory variations in perfusion index, has been shown to predict fluid responsiveness in mechanically ventilated patients; however, vasomotor tone changes induced by hypercapnia may affect PI and therefore reduce the accuracy of PVI.

Artificial pneumoperitoneum, which is commonly used in laparoscopic procedures and created with the Trendelenburg position and CO2 (carbon dioxide) insufflation, frequently leads to physiological changes such as PONV (postoperative nausea and vomiting) and pain. Although the mechanisms underlying its development are still unclear, PONV is caused by dopamine and serotonin released as a result of ischemia in the brain and intestinal tract, stimulating the medullary vomiting center. Therefore, ischemia has been shown to be one of the important factors for PONV. Hypocapnia is known to be associated with decreased cardiac output, and increased systematic vascular resistance can reduce blood flow in the brain and intestinal tract. Therefore, this study concluded that intraoperative hypocapnia may increase the risk of PONV. Another study reported that CO2 is a strong vasodilator and that intraoperative hypercarbia may be associated with increased perfusion to regions effective for PONV, including the brain and gastrointestinal tract. In a study examining the relationship between PI and postoperative pain, it was stated that there was a decrease in PI due to the activation of the sympathetic nervous system by pain, contraction in peripheral blood vessels and an increase in vasomotor tone, and an increase in PI values after the use of analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Planned for elective total laparoscopic hysterectomy
* 20-65 years old
* ASA I - II

Exclusion Criteria:

* history of intracranial disease
* lung disease
* systemic hypertension
* ischemic heart disease
* history of postoperative nausea and vomiting in previous operations
* smoking habit
* motion sickness
* liver and kidney dysfunction
* abnormal fluid-electrolyte balance
* preoperative use of antiemetic drugs
* severe heart failure
* ASA III and above
* body mass index> 35 kg m2

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective, randomized, controlled study was initiated at Kanuni Sultan Süleyman E.A.H. to measure the carbon dioxide changes that develop during laparoscopic operations with non-invasive monitoring, to evaluate the correlation between them, and to investigate their effects on postoperative pain and nausea and vomiting.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Investigation of the incidence of postoperative nausea, vomiting and pain | From enrollment to postoperative 1st week

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi Kanuni Sultan Süleyman Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)